CLINICAL TRIAL: NCT00557323
Title: A Long-term, Observational Study to Monitor Mortality, Bone-related Adverse Events and the Safety of Subjects Who Were Recruited Into Study SPD405-309
Brief Title: Long-term Effect of Lanthanum Carbonate on Bone
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SPD405-402
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Results first posted 2011-06-15 (Estimated); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia | interventions — lanthanum carbonate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients being treated for hyperphosphatemia with any marketed product
  Interventions: Drug: Lanthanum carbonate

INTERVENTIONS:
Drug: Lanthanum carbonate

SUMMARY:
Patients enrolled in a previous study (SPD405-309), who were exposed to lanthanum carbonate (Fosrenol), were eligible to continue on any prescribed treatment for hyperphosphatemia, including lanthanum carbonate (Fosrenol), for an additional 5 years. Patients were being observed for any bone adverse events or other serious adverse events, as well as the collection of mortality data.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who had exposure to lanthanum carbonate in SPD405-309

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patients from study SPD405-309 who were exposed to lanthanum carbonate
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2007-03-15 (Actual); Primary Completion 2010-08-31 (Actual); Study Completion 2010-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (19):
- United States (8):
  - Imperial care Dialysis Center, Lynwood, California
  - Barnett Research and Communications Medical Group, Torrance, California
  - Western new England Renal & Transplant Associates, Springfield, Massachusetts
  - Mercy Medical Center, Canton, Ohio
  - Hypertension & Nephrology, Inc., Providence, Rhode Island
  - Nephrology Associates, PC, Nashville, Tennessee
  - University of Vermont, Burlington, Vermont
  - Nephrology Associates, PC, Richmond, Virginia
- Germany (8):
  - Bad König, Hesse
  - KfH Zentrum, Aachen
  - Dialysenzentrum, Bad Homburg
  - KfH Kuratorium duer Dialyse und Nierentransplanta Dialysezentrum Moabit, Berlin
  - KfH Dialysezentrum, Berlin
  - Dialysezentrum Barmbek, Hamburg
  - Dialysepraxis Altona, Hamburg
  - KfH Dialysezentrum, Rosenheim
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge
  - St. Helier Hospital, Carshalton
  - Manchester Royal Infirmary, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Followed subjects from study SPD405-309 (NCT00150540) for 5 years.
Groups:
- 5-Year Observational Period: Followed subjects previously exposed to lanthanum carbonate in study SPD405-309 (NCT00150540). Subjects were not issued investigational medicinal product. Subjects could be treated for hyperphosphatemia as prescribed by their physician during the study, although this was not required for participation. Treatment was not restricted by the protocol, and it could include treatment with lanthanum carbonate or any other phosphate binder as prescribed by the treating physician. Subjects were assessed every 6 months throughout the 5-year observational period. Data were collected on bone-related adverse events, serious adverse events and deaths.
Period: Overall Study
Arm/Group | 5-Year Observational Period
Started | 34
Completed | 27
Not Completed | 7
Not completed — Death | 3
Not completed — Withdrawal by Subject | 2
Not completed — Administrative change | 2

BASELINE CHARACTERISTICS:
Arm/Group | 5-Year Observational Period
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.1 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
  Germany | 18
  United Kingdom | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Study-emergent Bone-related Adverse Events (AEs)
Time Frame: 5 years
Population: Safety Set defined as all subjects who received at least one safety measurement during the study.
Measure: Number; unit: Bone-related AEs
Arm/Group | 5-Year Observational Period
Number analyzed (Participants) | 34
Bone-related AEs
  Fracture (8 subjects) | 9
  Arthralgia (1 subject) | 2
  Hyperparathyroidism tertiary | 1
  Flat feet | 1
  Fracture nonunion | 1
  Intervertebral disc protrusion | 1
  Osteoarthritis | 1
  Osteonecrosis | 1
  Osteopenia | 1
  Osteoporosis | 1
  Pain in extremity | 1
  Renal osteodystrophy | 1
  Tendonitis | 1

2. Secondary Outcome: Number of Study-emergent Deaths
Time Frame: 5 years
Population: Safety Set
Measure: Number; unit: Participants
Arm/Group | 5-Year Observational Period
Number analyzed (Participants) | 34
Participants | 3

ADVERSE EVENTS:
Description: Safety Set
Arm/Group | 5-Year Observational Period
Serious Adverse Events (participants affected / at risk) | 18/34
Other Adverse Events (participants affected / at risk) | 5/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-Year Observational Period (N=34)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Hyperparathyroidism tertiary (Endocrine disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Bronchitis acute (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 2 (2)
Pacemaker complication (Injury, poisoning and procedural complications) | 1 (1)
Shunt stenosis (Injury, poisoning and procedural complications) | 1 (1)
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 (3)
Subdural hematoma (Injury, poisoning and procedural complications) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (2)
Ureteric stenosis (Renal and urinary disorders) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Aneurysm arteriovenous (Vascular disorders) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 1 (1)
Peripheral occlusive disease (Vascular disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-Year Observational Period (N=34)
Fracture (Musculoskeletal and connective tissue disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.